CLINICAL TRIAL: NCT03237819
Title: Interest of Magnesium Sulfate in Thrombotic Thrombocytopenic Purpura in Intensive Care: Multicentric Randomized Controlled Trial
Brief Title: Magnesium Sulfate in Thrombotic Thrombocytopenic Purpura in Intensive Care
Acronym: MAGMAT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AOR16028
Record Dates: First submitted 2017-06-13; First posted 2017-08-03 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-06

CONDITIONS: Thrombotic Thrombocytopenic Purpura
Keywords: Thrombotic Thrombocytopenic Purpura; Intensive care
MeSH Terms: conditions — Purpura, Thrombotic Thrombocytopenic | interventions — Magnesium Sulfate

STUDY DESIGN:
Intervention Model Description: multicentre double-blind randomized clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: For each day of treatment, 4 ampoules of 10 ml will be distributed to the patient's nurse (4 ampoules of 1.5g of magnesium sulphate or 3 ampoules of 5% glucose as placebo).
  The bulbs will be labeled identically so that the blind can be maintained Moreover, in order to preserve the blind, the dosage of magnesemia should not be performed outside of a necessity judged by the clinician in charge of the patient
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Glucose serum (3 ampoules)
  Interventions: Drug: Placebo - Concentrate
- Magnesium Sulfate (Experimental): 20/5000 magnesium sulfate (4 ampoules, 1,5g each)
  Interventions: Drug: Sulfate, Magnesium

INTERVENTIONS:
Drug: Sulfate, Magnesium — Magnesium sulphate will be administered at a dose of 6g over 20 min intravenously followed by a continuous infusion of 6g / 24h for 3 days.
  For each day of treatment, 4 ampoules of 10 ml will be distributed to the nurse in charge of the patient (4 ampoules of 1,5g of magnesium sulfate)
  Arms: Magnesium Sulfate
Drug: Placebo - Concentrate — For each day of treatment, 4 ampoules of 10 ml will be distributed to the nurse in charge of the patient (4 ampoules of glucose 5% as placebo)
  Arms: Placebo

SUMMARY:
Thrombotic Thrombocytopenic Purpura (TTP) is a potentially life-threatening thrombotic microangiopathy caused by a severe deficiency of ADAMTS13 (a disintegrin and metalloproteinase with a thrombospondin type 1 motif member 13). Decreased ADAMTS13 activity leads to an accumulation of ultralarge von Willebrand factor (vWF) multimers which induce aggregation of platelets and microthrombi. These microthrombi may involve the brain, heart, kidneys and lead to life-threatening organ failures.

In experimental models, magnesium sulfate increases cleavage of newly released vWF by ADAMTS13, decreases the endothelial secretion of ultralarge vWF and inhibits the interaction of vWF with platelets. In another thrombotic microangiopathy, magnesium sulfate has been shown to reduce the risk of seizures in women with severe pre-eclampsia. In analogy with its evidence-based therapeutic application in pre-eclampsia and based on a strong rationale for magnesium supplementation in TTP, we propose a phase 3, double blind, placebo controlled, and randomized study to evaluate the efficacy of magnesium sulfate in more rapidly restoring normal platelet counts as measure of prevention of further microvascular thrombosis in patients with Thrombotic Thrombocytopenic Purpura.

ELIGIBILITY:
Inclusion Criteria:

* Age > or = 18 years
* Health insurance
* Signed inform consent by patient or relatives

Exclusion Criteria:

* Pregnancy
* No health insurance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2018-05-27 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Time to normalization of the platelet count | 3 months
  Normalization of the platelet is defined as a platelet count that reaches at least 150,000 per cubic millimeter for 48 consecutive hours

SECONDARY OUTCOMES:
Duration and volume of plasma exchanges | 30 days
platelet count | 5 days
proportion of subjects with refractory TTP | 5 days
  absence of platelet count doubling after 4 days of standard treatment
Proportion of subjects with an exacerbation of TTP | 30 days
  recurrence during the 30 days after the last daily plasma exchange
Proportion of subjects with a relapse of TTP | 3 months
  recurrence occurring more than 30 days after the last daily plasma exchange
Cardiac trouble frequency | day 30
Cerebral trouble frequency | day 30
Acute kidney injury | day 30
  Kidney Disease: Improving Global Outcomes (KDIGO) score > or = 1
Time to normalization of hemolysis marker levels | day 30
  Lactate dehydrogenase (LDH), haptoglobin, bilirubinemia, hemoglobin
Hospital length of stay | day 90
Hospital mortality | day 90
  90 days after randomization
ICU length of stay | day 90
ICU mortality | day 90
Adverse events related to the use of magnesium sulfate | day 7

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Louis hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided